CLINICAL TRIAL: NCT05576558
Title: The Effect of Occupational Therapy on Anxiety, Depression, and Psychological Well-Being Symptoms in the Elderly: A Single-Blind Randomized-Controlled Study
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, SEDA DEĞİRMENCİ ÖZ, Assist.Prof.Dr., Istanbul Aydın University
Other Study IDs: Istanbul AU
Record Dates: First submitted 2022-09-29; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: The Effect of Occupational Therapy on Anxiety, Depression, and Psychological Well-Being Symptoms in the Elderly
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Participants were assigned to intervention and control groups according to the randomization list previously prepared by the researchers. All participants were first informed about the study and their informed consent was obtained. Participant Information Form, Geriatric Anxiety Scale, Psychological Well-Being Scale, and Geriatric Depression Scale were filled out by all participants.

The elderly in the intervention group were divided into 5 groups of 10 and a time was determined for the session in cooperation with the participants in each subgroup. A 60-minute therapy session was administered by the occupational expert. The applications were carried out in a total of 7 sessions as a daily session. The control group was not subjected to any application. Geriatric Anxiety Scale, Psychological Well-Being Scale, and Geriatric Depression Scale were refilled for the second time in all elderly on the 7th day after the application.

DETAILED DESCRIPTION:
Participants were assigned to intervention and control groups according to the randomization list previously prepared by the researchers. All participants were first informed about the study and their informed consent was obtained. Participant Information Form, Geriatric Anxiety Scale, Psychological Well-Being Scale, and Geriatric Depression Scale were filled out by all participants.

The elderly in the intervention group were divided into 5 groups of 10 and a time was determined for the session in cooperation with the participants in each subgroup. A 60-minute therapy session was administered by the occupational expert. The applications were carried out in a total of 7 sessions as a daily session. The control group was not subjected to any application. Geriatric Anxiety Scale, Psychological Well-Being Scale, and Geriatric Depression Scale were refilled for the second time in all elderly on the 7th day after the application.

ELIGIBILITY:
Inclusion Criteria:

* The elderly, who agreed to participate in the study,
* were aged 60 and over, were cooperative,
* had no communication problems,
* and did not receive any training, course, or practice on coping with anxiety, tension, and stress were included in the sample.

Exclusion Criteria:

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study was carried out between April and August 2022 with the elderly living in a private elderly care center in Istanbul/Turkey.
  The elderly, who agreed to participate in the study, were aged 60 and over, were cooperative, had no communication problems, and did not receive any training, course, or practice on coping with anxiety, tension, and stress were included in the sample.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-08-26 (Actual); Study Completion 2022-09-19 (Actual)

PRIMARY OUTCOMES:
Participant Information Form | From April to August 2022
  It was created in line with the literature. It is a form containing sociodemographic data such as age, gender, educational status, etc.
Geriatric Anxiety Scale: | From April to August 2022
  It is a measurement tool that consists of 28 items and provides self-anxiety reporting of the elderly. The scale was developed by Pachana et al. (Pachana et al., 2007), and adapted to the Turkish language by Karahan et al. (Karahan et al., 2018). Participants were asked to indicate how often they experienced each symptom during the week including today. The response format uses a 4-point Likert scale ranging from 0 (never) to 3 (always), with higher scores indicating higher levels of anxiety. The scale covers three different subscales common among older adults. These are somatic (physical) subscale, 1, 6, 7, 15, 19, 20, 21 (7 items), cognitive symptoms 2, 3, 10, 14, 16, 17, 22, 23 (8 items), and mood subscale, 4, 5, 8, 9, 11, 12, 13, 18 (8 items). The GAS total score is based on the first 23 items. Since items 24-28 are used by clinicians to determine the area of anxiety, they are not used in total scoring.
Psychological Well-Being Scale | From April to August 2022
  The scale developed by Diener, Scollon, & Lucas, (2009) to measure the level of psychological well-being has eight items. It identifies important elements of human function, including positive relationships, feeling of efficacy, and having a meaningful and purposeful life. The Turkish validity and reliability of the scale were made by Telef in 2013. Scale items are scored between 1 (strongly disagree) and 7 (strongly agree). All items are structured positively. Scores range from 8 (strongly disagree with all items) to 56 (strongly agree with all items). A high score on the scale indicates a high psychological strength of the individual.
Geriatric Depression Scale | From April to August 2022
  It was developed by Yesavage to evaluate the depressive symptoms of elderly individuals and consists of a total of 15 questions (Yesavage & Sheikh, 1986). It is designed in such a way that the elderly can mark it easily and can be answered as "yes" or "no". Items 1, 5, 7, 11, and 13 in the scale are structured positively, while other items are structured negatively. In the scoring of the scale, 1 point is given for each response in favor of depression and 0 points for other responses. A score of "5 and above" on the scale is considered a significant finding for the diagnosis of depression (Akturk, Sahin, Dagdeviren & Ozer, 2002).

CONTACTS AND LOCATIONS:
Overall Officials: SEDA DEĞİRMENCİ ÖZ, Dr., Study Chair — Istanbul Aydın University
Locations (1):
- Seda Değirmenci Öz, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Degirmenci Oz S, Sezer E, Yildirim D. The effect of occupational therapy on anxiety, depression, and psychological well-being in older adults: a single-blind randomized-controlled study. Eur Geriatr Med. 2024 Feb;15(1):217-223. doi: 10.1007/s41999-023-00900-z. Epub 2023 Dec 16. PMID 38103144